CLINICAL TRIAL: NCT03547921
Title: Primary Upper Limb Deep Vein Thrombosis. Is First Rib Resection Necessary?
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Sheba Medical Center (Other Government)
Responsible Party: Principal Investigator, Dr. Daniel Silverberg, vascular surgeon, Sheba Medical Center
Other Study IDs: sheba-18-4765-DS-CTIL
Record Dates: First submitted 2018-03-28; First posted 2018-06-06 (Actual); Last update posted 2018-06-06 (Actual); Status verified 2018-05

CONDITIONS: Paget Schroetter Syndrome
MeSH Terms: conditions — Upper Extremity Deep Vein Thrombosis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- operative: operative
  Interventions: Device: iu22 ultrasound system - phillips
- non operative: non operative
  Interventions: Device: iu22 ultrasound system - phillips

INTERVENTIONS:
Device: iu22 ultrasound system - phillips — iu22 ultrasound system - phillips

SUMMARY:
The purpose of the study is to compare outcome of patients with effort thrombosis who were treated operatively to those treated nonoperatively

ELIGIBILITY:
Inclusion Criteria:\

* patients treated for upper extremity DVT

Exclusion Criteria:

* none

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: patients who were previously treated for upper extremity DVT ( anticoagulation- with or without 1st rib resection)
Sampling Method: Non-Probability Sample
Enrollment: 20 (Estimated)
Dates: Start 2018-07-01 (Estimated); Primary Completion 2018-07-01 (Estimated); Study Completion 2018-09-01 (Estimated)

PRIMARY OUTCOMES:
clinical differences | 10years
  clinical differences between the 2 groups Patients will be evaluated by the " Villata" post thrombotic syndrome (PTS) scoring system. The sum of each parameter will be used to compare he groups Vilata PTS scoring system: ( 0- ABSENT , 3 SEVERE ) Symptoms/clinical signs None Mild Moderate Severe Symptoms Pain Cramps Heaviness Pruritus Clinical signs edema Skin induration Hyperpigmentation Redness Venous ectasia Pain on calf compression

SECONDARY OUTCOMES:
vein patency | 10 years
  patency of SCV based on duplex